CLINICAL TRIAL: NCT01921205
Title: A Multicenter, Double Blind, Randomized, Placebo Controlled, Parallel Group Study to Investigate the Efficacy and Safety of Lacosamide as Adjunctive Therapy in Subjects With Epilepsy ≥4 Years to <17 Years of Age With Partial Onset Seizures
Brief Title: Study to Investigate Lacosamide as Add-on Therapy in Subjects ≥4 Years to <17 Years of Age With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP0969; 2012-004996-38 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; UCB; Epilepsy; Partial Onset Seizures; Pediatric
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lacosamide (Experimental)
  Interventions: Drug: Lacosamide
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lacosamide — Subjects <30 kg (LCM oral solution): 4 mg/kg - 6 mg/kg BID ( 8mg/kg/day - 12 mg/kg/day)
  Subjects ≥30 kg to <50 kg (LCM oral solution): 3 mg/kg - 4 mg/kg BID (6 mg/kg/day - 8 mg/kg/day)
  Subjects ≥50 kg (LCM tablets): 150 mg - 200 mg BID (300 mg/day - 400 mg/day)
  Other Names: Vimpat(R)
  Arms: Lacosamide
Other: Placebo — Subjects <30 kg (placebo oral solution): 4 mg/kg - 6 mg/kg BID (8 mg/kg/day - 12 mg/kg/day)
  Subjects ≥30 kg to <50 kg (placebo oral solution): 3 mg/kg - 4 mg/kg BID (6 mg/kg/day - 8 mg/kg/day)
  Subjects ≥50 kg (placebo tablets): 150 mg - 200 mg BID (300 mg/day - 400 mg/day)
  Arms: Placebo

SUMMARY:
Study to evaluate the efficacy of Lacosamide (LCM) administered in addition to 1 to ≤3 other Anti-Epileptic Drugs in subjects with epilepsy ≥4 years to <17 years of age who currently have uncontrolled partial onset seizures.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of LCM administered concomitantly with 1 to ≤3 Anti-Epileptic Drugs (AEDs) in subjects with epilepsy ≥4 years to <17 years of age who currently have uncontrolled partial onset seizures.

The secondary objective is to evaluate the safety and tolerability of LCM in subjects ≥4 years to <17 years of age.

An additional objective is to evaluate the pharmacokinetics (PK) of LCM in subjects ≥4 years to <17 years of age.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form is signed and dated by the parent(s) or legal representative. The Informed Consent form or a specific Assent form, where required, will be signed and dated by minors
* Subject/legal representative is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, and medication intake according to the judgment of the investigator
* Subject is male or female from ≥4 years to <17 years of age
* Subject has a diagnosis of Epilepsy with partial-onset seizures. The results of ≥1 prior electroencephalogram (EEG) AND 1 prior magnetic resonance imaging/computerized tomography scan should be consistent with the above diagnosis
* Subject has been observed to have uncontrolled partial-onset seizures after an adequate course of treatment (in the opinion of the investigator) with ≥2 Anti-Epileptic Drugs (AEDs) (concurrently or sequentially)
* Subject must have been observed to have on average ≥2 partial onset seizures per 28 days with seizure free phase no longer than 21 days in the 8 week period prior to entry into the Baseline Period. During this study, subjects must have reported ≥2 partial onset seizures during the 8 week prospective Baseline Period to be eligible for randomization at Visit 2. (Note: In the case of simple partial onset seizures, only those seizures with motor signs will be counted towards meeting the inclusion criterion.)
* Subject is on a stable dosage regimen of 1 to ≤3 AEDs. The daily dosage regimen of concomitant AED therapy must be kept constant for a period of ≥4 weeks prior to the Baseline Period
* Vagal nerve stimulation (VNS) is allowed and will not be counted as a concomitant AED. The VNS device must be implanted for ≥6 months before Visit 1, and the device settings must be stable for ≥4 weeks before Visit 1 and be kept stable during the Baseline Period. Use of the VNS device magnet is allowed

Exclusion Criteria:

* Subject has previously participated in this study or subject has been assigned to Lacosamide (LCM) in a previous LCM study
* Subject has participated in another study of an investigational medicinal product (IMP) or a medical device within ≤2 months of Visit 1 or is currently participating in another study of an IMP or a medical device
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject ≥6 years of age has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C SSRS) at Screening
* Subject has a known hypersensitivity to any component of the IMP or has ever received LCM
* Female subject who is pregnant or nursing, and/or a female subject of childbearing potential who is not surgically sterile or does not practice 1 highly effective method of contraception (according to International Conference on Harmonisation [ICH] guidance defined as those that result in a failure rate of less than 1% per year when used consistently and correctly), unless sexually abstinent, for the duration of the study. Female subject of childbearing potential taking enzyme inducing antiepileptic drugs (EI AEDs: carbamazepine, phenytoin, barbiturates, primidone, topiramate, oxcarbazepine) who is not surgically sterile or does not practice 1 highly effective method of contraception according to the WHO recommendation (ie, depot medroxyprogesterone acetate, norethisterone enantate, intrauterine devices, combined injectables, and progestogen implants) with administration of EI AEDs OR does not practice 2 combined methods of contraception (ie, combined hormonal contraception plus barrier method with spermicidal agent), unless sexually abstinent, for the duration of the study
* Subject has a medical condition that could be expected in the opinion of the investigator to interfere with drug absorption, distribution, metabolism, or excretion
* Subject has experienced febrile seizures exclusively. The occurrence of febrile seizures in addition to other unprovoked seizures is not exclusionary
* Subject is on a ketogenic or other specialized diet. If the subject was on a specialized diet in the past, they must be off the diet for ≥2 months prior to the Baseline Period
* Subject has an alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin level ≥2 times the upper limit of normal (ULN), or creatinine clearance less than 30 mL/min
* Subject has a clinically relevant ECG abnormality, in the opinion of the investigator (eg, second or third degree heart block at rest or a corrected QT interval [QTc] greater than 450 ms)
* Subject has hemodynamically significant congenital heart disease
* Subject has an arrhythmic heart condition requiring medical therapy
* Subject has a known history of severe anaphylactic reaction or serious blood dyscrasias
* Subject has nonepileptic events that could be confused with seizures
* Subject has a current diagnosis of Lennox-Gastaut syndrome, primary generalized epilepsy, mixed seizure disorder (partial and primarily generalized seizures), or purely nocturnal seizures
* Subject has a history of convulsive status epilepticus ≤2 months prior to the Baseline Period
* Subject has been treated with vigabatrin and experienced any vision loss. Subjects who have received vigabatrin in the past must have documentation of an assessment for vision loss prior to study entry or documentation of why visual field testing cannot be performed
* Subject has been treated with felbamate and has experienced any serious toxicity issues (defined as liver failure, aplastic anemia) with this treatment. Subjects treated with felbamate for <12 months are excluded. Note: any subject who has been treated with felbamate for ≥12 months and has not experienced serious toxicity issues is eligible
* Subject has a medically documented history of alcohol or drug abuse
* Subject has a known cardiac sodium channelopathy, such as Brugada syndrome
* Subject has an acute or sub acutely progressive central nervous system disease. Subject has epilepsy secondary to a progressing cerebral disease or any other progressively neurodegenerative disease (malignant brain tumor or Rasmussen Syndrome)

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2013-08-29; Primary Completion 2017-01-24 (Actual); Study Completion 2017-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493
Locations (118):
- United States (13):
  - 127, Boulder, Colorado
  - 105, Orlando, Florida
  - 117, Tampa, Florida
  - 103, Atlanta, Georgia
  - 124, Lexington, Kentucky
  - 112, Louisville, Kentucky
  - 121, Shreveport, Louisiana
  - 115, Las Vegas, Nevada
  - 102, Charlotte, North Carolina
  - 640, Eugene, Oregon
  - 122, Dallas, Texas
  - 101, Tomball, Texas
  - 114, Seattle, Washington
- Argentina (2):
  - 143, Buenos Aires
  - 142, Córdoba
- Australia (3):
  - 200, Heidelberg West
  - 203, Herston
  - 205, South Brisbane
- 304, Brussels, Belgium
- Bulgaria (2):
  - 310, Sofia
  - 312, Sofia
- Colombia (2):
  - 172, Floridablanca
  - 171, Medellín
- Croatia (3):
  - 613, Osijek
  - 610, Rijeka
  - 612, Zagreb
- Czechia (4):
  - 321, Hradec Králové
  - 320, Ostrava-Poruba
  - 322, Prague
  - 323, Prague
- Estonia (2):
  - 331, Tallinn
  - 330, Tartu
- Georgia (4):
  - 620, Tbilisi
  - 621, Tbilisi
  - 622, Tbilisi
  - 623, Tbilisi
- Hungary (7):
  - 361, Budapest
  - 362, Budapest
  - 363, Budapest
  - 364, Budapest
  - 360, Debrecen
  - 367, Miskolc
  - 366, Pécs
- Israel (4):
  - 370, Holon
  - 371, Kfar Saba
  - 374, Petah Tikva
  - 372, Tel Aviv
- Italy (9):
  - 384, Bologna
  - 388, Florence
  - 387, Genova
  - 380, Mantova
  - 381, Milan
  - 393, Padua
  - 383, Roma
  - 392, Roma
  - 386, Verona
- Latvia (2):
  - 400, Riga
  - 402, Valmiera
- 411, Kaunas, Lithuania
- Mexico (3):
  - 569, Culiacán
  - 563, Guadalajara
  - 568, Monterrey
- 660, Podgorica, Montenegro
- Poland (11):
  - 433, Gdansk
  - 432, Katowice
  - 420, Kielce
  - 422, Krakow
  - 431, Krakow
  - 423, Poznan
  - 425, Poznan
  - 421, Szczecin
  - 429, Tyniec Mały
  - 430, Warsaw
  - 428, Wroclaw
- Romania (6):
  - 574, Bucharest
  - 572, Cluj-Napoca
  - 576, Sibiu
  - 580, Suceava
  - 570, Timișoara
  - 577, Timișoara
- Russia (8):
  - 443, Kazan'
  - 444, Kazan'
  - 442, Moscow
  - 449, Moscow
  - 441, Saint Petersburg
  - 446, Saint Petersburg
  - 440, Smolensk
  - 447, Voronezh
- Serbia (5):
  - 464, Belgrade
  - 460, Kragujevac
  - 461, New Belgrade
  - 462, Novi Sad
  - 463, Novi Sad
- Slovakia (3):
  - 470, Bardejov
  - 473, Nitra
  - 472, Nové Zámky
- 670, Ljubljana, Slovenia
- South Korea (5):
  - 211, Daegu
  - 210, Seoul
  - 212, Seoul
  - 213, Seoul
  - 215, Seoul
- Taiwan (3):
  - 220, Changhua
  - 222, Taichung
  - 224, Taipei
- Thailand (6):
  - 232, Bangkok
  - 236, Bangkoknoi
  - 231, Muang
  - 233, Muang
  - 235, Pathumwan
  - 230, Ratchathewi
- Ukraine (4):
  - 602, Dnipropetrovsk
  - 606, Kiev
  - 682, Uzhhorod
  - 603, Vinnitsa
- United Kingdom (3):
  - 514, Birmingham
  - 515, Birmingham
  - 511, Leeds

REFERENCES:
- [Derived] Johnson ME, McClung C, Bozorg AM. Analyses of seizure responses supportive of a novel trial design to assess efficacy of antiepileptic drugs in infants and young children with epilepsy: Post hoc analyses of pediatric levetiracetam and lacosamide trials. Epilepsia Open. 2021 Jun;6(2):359-368. doi: 10.1002/epi4.12482. Epub 2021 May 3. PMID 34033237
- [Derived] Babar RK, Bresnahan R, Gillespie CS, Michael BD. Lacosamide add-on therapy for focal epilepsy. Cochrane Database Syst Rev. 2021 May 17;5(5):CD008841. doi: 10.1002/14651858.CD008841.pub3. PMID 33998660
- [Derived] Farkas V, Steinborn B, Flamini JR, Zhang Y, Yuen N, Borghs S, Bozorg A, Daniels T, Martin P, Carney HC, Dimova S, Scheffer IE; SP0969 Study Group. Efficacy and tolerability of adjunctive lacosamide in pediatric patients with focal seizures. Neurology. 2019 Sep 17;93(12):e1212-e1226. doi: 10.1212/WNL.0000000000008126. Epub 2019 Aug 28. PMID 31462582
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in August 2013 and concluded in January 2017.
Pre-assignment Details: The Participant Flow refers to the Safety Set which included all randomized subjects who took at least 1 dose of study medication.
Groups:
- Placebo: This arm includes subjects with epilepsy, who received a flexible dose of Placebo oral solution or tablets, administered twice a day. Appearance of Placebo oral solution and tablets matched the Lacosamide oral solution and tablets.
- Lacosamide: This arm includes subjects with epilepsy, who received a flexible dose of Lacosamide (LCM) oral solution or tablets, administered twice a day. Subjects weighing <30kg received 8mg/kg/day to 12mg/kg/day Lacosamide (LCM) oral solution; subjects weighing >=30kg to <50kg received 6mg/kg/day to 8mg/kg/day LCM oral solution; and subjects weighing >=50kg received 300mg/day to 400mg/day LCM tablets, or if unable or unwilling to swallow tablets may have received LCM oral solution, however, they were not permitted to exceed the maximum dose of LCM 400mg/day. The subject's body weight at Baseline (Visit 2) was used to determine the dose throughout the study.
Period: Overall Study
Arm/Group | Placebo | Lacosamide
Started | 172 | 171
Completed | 151 | 151
Not Completed | 21 | 20
Not completed — Adverse Event | 12 | 7
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Use Of Prohibited Medication | 0 | 1
Not completed — The Excessive Use Of Rescue Medication | 0 | 1
Not completed — Non Compliance Of The Parent | 0 | 1
Not completed — Non Compliance Of Child | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics refers to the Safety Set which included all randomized subjects who took at least 1 dose of study medication.
Arm/Group | Placebo | Lacosamide | Total Title
Number analyzed (Participants) | 172 | 171 | 343
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 172 | 171 | 343
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (3.5) | 10.5 (3.6) | 10.7 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 80 | 153
  Male | 99 | 91 | 190
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 35 | 25 | 60
  Black or African American | 1 | 2 | 3
  White | 129 | 138 | 267
  Other/Mixed | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Partial Onset Seizure (POS) Frequency Per 28 Days From Baseline to the Maintenance Period
Description: The POS frequency is standardized to a 28-day duration. Negative values indicate improvement from Baseline.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: The analysis was performed on the Full Analysis Set (FAS), which included all subjects who were randomized, received at least 1 dose of study medication, and had a Baseline and at least 1 post-Baseline assessment of seizure frequency data. Only subjects with available data were included in this analysis.
Measure: Median (Full Range); unit: Seizures per 28 days
Groups:
- Placebo (FAS): This arm includes subjects with epilepsy, who received a flexible dose of Placebo oral solution or tablets, administered twice a day. Appearance of Placebo oral solution and tablets matched the Lacosamide oral solution and tablets.
- Lacosamide (FAS): This arm includes subjects with epilepsy, who received a flexible dose of Lacosamide (LCM) oral solution or tablets, administered twice a day. Subjects weighing <30kg received 8mg/kg/day to 12mg/kg/day Lacosamide (LCM) oral solution; subjects weighing >=30kg to <50kg received 6mg/kg/day to 8mg/kg/day LCM oral solution; and subjects weighing >=50kg received 300mg/day to 400mg/day LCM tablets, or if unable or unwilling to swallow tablets may have received LCM oral solution, however, they were not permitted to exceed the maximum dose of LCM 400mg/day. The subject's body weight at Baseline (Visit 2) was used to determine the dose throughout the study.
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 168 | 170
Seizures per 28 days | -1.55 [-318.7 to 690.0] | -3.05 [-302.9 to 210.4]
Statistical Analysis 1: Comparison: Placebo (FAS) vs Lacosamide (FAS); Test type: Superiority; p = 0.0003, ANCOVA; Seizure frequency (log transformed) is analyzed using analysis of covariance with terms for treatment, pooled center and Baseline seizure frequency; Percent reduction over Placebo = 31.72, 95% CI 2-sided [16.342 to 44.277] — Percent reduction over placebo is estimated as 100 x (1-exp[LSMLacosamide-LSMPlacebo]). Where LSM is Least Square Mean

2. Secondary Outcome: Proportion of Responders Where a Responder is Defined as a Participant With >= 50% Reduction in Partial Onset Seizure Frequency Per 28 Days From Baseline to the Maintenance Period
Description: Proportion of responders is presented as percentage of participants. A responder is a subject experiencing a 50 % or greater reduction in partial onset seizure frequency per 28 days from Baseline to the Maintenance Period.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: The analysis was performed on the Full Analysis Set (FAS), which included all subjects who were randomized, received at least 1 dose of study medication, and had a Baseline and at least 1 post-Baseline assessment of seizure frequency data. Only subjects with response data have been included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 168 | 170
percentage of participants | 33.3 | 52.9

3. Secondary Outcome: Proportion of Subjects Experiencing a >=25 % to <50 %, 50 % to 75 %, or >75 % Reduction in Partial Onset Seizure Frequency Per 28 Days From Baseline to the End of Maintenance Period
Description: Proportion of subjects is presented as percentage of participants. A >=25%-<50% response in the Maintenance Period is defined as >=25% to <50% reduction in POS frequency per 28 days from Baseline to end of Maintenance Period. A >=50%-<=75% response in the Maintenance Period is defined as >=50% to <=75% reduction in POS frequency per 28 days from Baseline to end of Maintenance Period. A 75% response in the Maintenance Period is defined as >75% reduction in POS frequency per 28 days from Baseline to end of Maintenance Period.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: The analysis was performed on the Full Analysis Set (FAS), which included all subjects who were randomized, received at least 1 dose of study medication, and had a Baseline and at least 1 post-Baseline assessment of seizure frequency data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 170 | 170
percentage of participants
  >=25% - <50% | 14.7 | 11.8
  >=50% - <=75% | 17.1 | 21.8
  >75% | 15.9 | 31.2

4. Secondary Outcome: Change in Partial Onset Seizure Frequency Per 28 Days From Baseline to the Entire Treatment (ie, Titration+Maintenance Periods)
Description: The POS frequency is standardized to a 28-day duration. Negative values indicate improvement from Baseline.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: as for outcome 1
Measure: Median (Full Range); unit: Seizures per 28 days
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 169 | 170
Seizures per 28 days | -1.22 [-250.6 to 477.0] | -2.46 [-219.2 to 210.4]

5. Secondary Outcome: Proportion of Subjects Experiencing a >=25 % to <50 %, 50 % to 75 %, or >75 % Reduction in Partial Onset Seizure Frequency Per 28 Days From Baseline to the Entire Treatment (ie, Titration+Maintenance Periods)
Description: Proportion of subjects is presented as percentage of participants. A >=25%-<50% response in the Treatment Period is defined as >=25% to <50% reduction in POS frequency per 28 days from Baseline to end of Treatment Period. A >=50%-<=75% response in the Treatment Period is defined as >=50% to <=75% reduction in POS frequency per 28 days from Baseline to end of Treatment Period. A 75% response in the Treatment Period is defined as >75% reduction in POS frequency per 28 days from Baseline to end of Treatment Period.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 170 | 170
percentage of participants
  >=25% - <50% | 15.3 | 16.5
  >=50% - <=75% | 20.6 | 20.6
  >75% | 8.8 | 23.5

6. Secondary Outcome: Proportion of Subjects Experiencing no Change in Partial Onset Seizure Frequency (Between <25 % Reduction and <25 % Increase) Per 28 Days From Baseline to the Entire Treatment (ie, Titration+Maintenance Periods)
Description: Proportion of subjects is presented as percentage of participants. No change is defined as between <25% reduction and <25% increase in POS frequency per 28 days from Baseline to the entire Treatment Period, otherwise not between <25% reduction and <25% increase is defined as a change.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 169 | 170
percentage of participants | 32.0 | 20.6

7. Secondary Outcome: Proportion of Subjects Experiencing an Increase in Partial Onset Seizure Frequency Per 28 Days of >=25 % From Baseline to the Entire Treatment (ie, Titration+Maintenance Periods)
Description: Proportion of subjects is presented as percentage of participants. An increase is defined as a >=25% increase in POS frequency per 28 days from Baseline to the entire Treatment Period, otherwise <25% increase is defined as no increase.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 169 | 170
percentage of participants | 23.1 | 18.8

8. Secondary Outcome: Change in Partial Onset Seizure Frequency Per 28 Days From Baseline to the Entire Treatment (ie, Titration+Maintenance Periods) for Simple Partial Seizures
Description: The POS frequency is standardized to a 28-day duration. Negative values indicate improvement from Baseline.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: The analysis was performed on the Full Analysis Set (FAS), which included all subjects who were randomized, received at least 1 dose of study medication, and had a Baseline and at least 1 post-Baseline assessment of seizure frequency data. Only subjects with Simple Partial Seizures were included in this analysis.
Measure: Median (Full Range); unit: Seizures per 28 days
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 68 | 77
Seizures per 28 days | -1.14 [-250.6 to 477.0] | -1.25 [-217.4 to 100.2]

9. Secondary Outcome: Change in Partial Onset Seizure Frequency Per 28 Days From Baseline to the Entire Treatment (ie, Titration+Maintenance Periods) for Complex Partial Seizures
Description: The POS frequency is standardized to a 28-day duration. Negative values indicate improvement from Baseline.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: The analysis was performed on the Full Analysis Set (FAS), which included all subjects who were randomized, received at least 1 dose of study medication, and had a Baseline and at least 1 post-Baseline assessment of seizure frequency data. Only subjects with Complex Partial Seizures were included in this analysis.
Measure: Median (Full Range); unit: Seizures per 28 days
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 99 | 109
Seizures per 28 days | -0.98 [-78.0 to 239.7] | -2.06 [-131.8 to 210.4]

10. Secondary Outcome: Change in Partial Onset Seizure Frequency Per 28 Days From Baseline to the Entire Treatment (ie, Titration+Maintenance Periods) for Secondary Generalized Seizures
Description: The POS frequency is standardized to a 28-day duration. Negative values indicate improvement from Baseline.
Time Frame: Baseline to Week 16 (or last value on treatment)
Population: The analysis was performed on the Full Analysis Set (FAS), which included all subjects who were randomized, received at least 1 dose of study medication, and had a Baseline and at least 1 post-Baseline assessment of seizure frequency data. Only subjects with Secondary Generalized Seizures were included in this analysis.
Measure: Median (Full Range); unit: Seizures per 28 days
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 69 | 63
Seizures per 28 days | -1.0 [-204.7 to 39.8] | -2.81 [-99.3 to 72.7]

11. Secondary Outcome: Proportion of Seizure Free Days During the Maintenance Period for Subjects Who Completed the Maintenance Period
Description: The proportion of seizure free days is calculated as (days with number of seizures = 0) divided by (days with recorded data in the subject diary), where 'days with recorded data in the subject diary' excludes any days where 'Not Done' is recorded.
Time Frame: Week 7 to Week 16
Population: Percentages are based on the number of subjects in the Full Analysis Set (FAS), which included all subjects who were randomized, received at least 1 dose of study medication, and had a Baseline and at least 1 post-Baseline assessment of seizure frequency data. Only subjects who completed the Maintenance Period have been included in this analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 154 | 152
days | 0.65 (0.35) | 0.71 (0.32)

12. Secondary Outcome: Proportion of Subjects Who Achieved "Seizure Free" Status (Yes/no) for Subjects Who Completed the Maintenance Period
Description: as for outcome 11
Time Frame: Week 7 to Week 16
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Lacosamide (FAS)
Number analyzed (Participants) | 154 | 152
percentage of participants | 9.7 | 15.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 1 until Safety Follow-Up Visit up to week 24.
Arm/Group | Placebo | Lacosamide
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/171
Serious Adverse Events (participants affected / at risk) | 13/172 | 11/171
Other Adverse Events (participants affected / at risk) | 61/172 | 85/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=172) | Lacosamide (N=171)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 4 (5) | 2 (2)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (4)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
Emotional disorder of childhood (Psychiatric disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=172) | Lacosamide (N=171)
Vomiting (Gastrointestinal disorders) | 11 (15) | 17 (22)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 8 (15)
Pyrexia (General disorders) | 10 (11) | 17 (21)
Nasopharyngitis (Infections and infestations) | 10 (10) | 20 (29)
Upper respiratory tract infection (Infections and infestations) | 10 (14) | 10 (13)
Pharyngitis (Infections and infestations) | 5 (5) | 10 (13)
Somnolence (Nervous system disorders) | 11 (14) | 28 (42)
Dizziness (Nervous system disorders) | 13 (14) | 18 (26)
Headache (Nervous system disorders) | 15 (25) | 14 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT01921205/SAP_000.pdf
  • Study Protocol (2015-03-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT01921205/Prot_001.pdf